CLINICAL TRIAL: NCT01985464
Title: Feasibility Study of Umbilical Cord Tissue Derived Mesenchymal Stem Cells (UC-MSC) in Disease Modifying Anti-Rheumatic Drugs (DMARD) Resistant Rheumatoid Arthritis
Brief Title: Umbilical Cord Tissue-derived Mesenchymal Stem Cells for Rheumatoid Arthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Translational Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBS-UCMSCRA-001
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2018-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; umbilical cord; mesenchymal; stem cells
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Umbilical cord mesenchymal stem cells (Experimental)
  Interventions: Biological: Umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Umbilical cord mesenchymal stem cells

SUMMARY:
Allogeneic human umbilical cord tissue-derived stem cells will be injected intravenously once per day for 5 days is a safe and useful procedure in inducing remission of RA in patients resistant to standard DMARD therapy.

DETAILED DESCRIPTION:
The proposed study will assess primarily safety and secondary efficacy endpoints of allogeneic UC-MSC administered to 20 patients with disease modifying antirheumatic drug (DMARD)-resistant Rheumatoid Arthritis (RA) who have been non-responsive to at least one course of one DMARD selected from a group comprising of: gold salts, leflunomide, methotrexate, and hydroxychloroquine.

The primary objective of safety will be defined as freedom from treatment associated adverse events for the period of one year. The secondary objective of efficacy will include evaluation at baseline and at months 3 and 12 of efficacy endpoints of C reactive protein (CRP), erythrocyte sedimentation rate (ESR), anti-citrulline antibody, rheumatoid factor (RF), Quality of Life Questionnaire, 28-joint disease activity score (DAS28), European League against Rheumatism (EULAR) response criteria and immunological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Signed inform consent by the subject.
* Age older than 18 years and ability to understand the planned treatment.
* Patients of either gender with RA with a duration of 6 months to 20 years defined as the presence of at least three of the following criteria: 3 or more painful, 2 or more swollen joints, morning stiffness for at least 45 minutes (on average during the week prior to entry), and an erythrocyte sedimentation rate (ESR) of at least 28 mm.
* Non-responsive to at least one course of one DMARD selected from the group comprising of: gold salts, leflunomide, methotrexate, and hydroxychloroquine.
* Second-line agents are discontinued at least 4 weeks prior to entry.
* Able to tolerate ALL study procedures
* Able to give informed Consent
* Negative for HcG with a serum pregnancy test
* Hematocrit ≥ 28.0%, White Blood Cell count ≤ 14,000, Platelet count ≥ 50,000,
* Life expectancy of 6 months or more in the opinion of the investigator
* Serum bilirubin, ALT, AST up to 2.5 time the upper level of normal.
* Controlled blood pressure (systolic blood pressure ≤140 and a diastolic blood pressure of ≤90 mmHG) and established anti-hypertensive therapy as necessary prior to entry into the study
* Patient has received stable, standard medical therapy for at least one month with no new medications to treat the disease introduced in the last month.
* Pre-existing condition (e.g. thromboembolic risk, diabetes, hypercholesterolemia) are adequately controlled in the opinion of the investigator
* Fertile patients (male and female) must agree to use an appropriate form of contraception while participating in the study.

Exclusion Criteria:

* Female who is pregnant or nursing, or of child-bearing potential and is not using a reliable birth control method, or who intend to become pregnant during the tenure of this study.
* History of prior radiation exposure for oncological treatment.
* History of Bone Marrow Disorder (especially NHL, MDS)
* History of abnormal bleeding or clotting.
* History of Liver Cirrhosis.
* End stage renal disease (Creatinine ≤ 3.0 mg / dl) and/or dialysis
* Active clinical infection being treated by antibiotics before one week enrollment
* Inability or unwillingness to comply with the treatment protocol, follow-up, research tests, or give consent.
* History of life-threatening arrhythmias, except if an automated implantable cardioverter defibrillator (AICD) is implanted
* Life expectancy <6 months due to concomitant illnesses
* Known cancer and undergoing treatment; chemotherapy and/or radiotherapy
* Patients receiving treatment with hematopoietic growth factors (e.g., EPO, G-CSF)
* Patients who can not stop anticoagulation therapy (warfarin) 72hrs prior to infusion
* Patients who can not stop anti-platelet therapy (clopidogrel) 7 days prior infusion
* Prior admission for substance abuse
* Body Mass Index (BMI) of 40 kg/m2 or greater
* Patient receiving experimental medication or participating in another clinical study within 30 days of signing the informed consent
* In the opinion of the investigator or the sponsor, the patient is unsuitable for cellular therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 12 months

SECONDARY OUTCOMES:
Number of participants with a change in disease activity index as measured by 28-DAS Score | 12 months
Number of participants with a change in current disease activity as measured by EULAR Response Criteria | 12 months
Change from baseline quality of life measure (based on Stanford HAQ) | 12 months
Change from baseline C-reactive protein | 12 months
Change from baseline erythrocyte sedimentation rate (ESR) | 12 months
Change from baseline anti-citrulline antibody measure | 12 months
Change from baseline rheumatoid factor (RF) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Castrellon, MD, Principal Investigator — Not Affiliated
Locations (1):
- Stem Cell Institute, Panama City, Panama